CLINICAL TRIAL: NCT06884553
Title: Effects of Robot-assistED Rehabilitation Versus OccupatIonal Therapy on the Functional Recovery of the Upper Limb in PatiEnts with Chronic STroke: a Randomized Controlled Trial
Brief Title: Robotic Rehabilitation Vs Occupational Therapy Chronic Stroke Upper Limb Rehabilitation
Acronym: REDIRECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Francesca Cecchi, Professor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REDIRECT
Record Dates: First submitted 2023-10-17; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Stroke
Keywords: Robotic rehabilitation; occupational therapy; chronic stroke; upper limb impairment; biomarkers; manual dexterity
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized controlled trial (RCT) designed for nonprofit purposes and aimed at demonstrating superiority.
Who Masked: Outcomes Assessor
Masking Description: The assessors conducting outcome evaluations and the operators performing statistical analysis will be blinded to the assignment group. Given the nature of the intervention, it will not be possible to maintain blinding regarding the treatment for both the therapists and the patients. To minimize bias related to patient non-blinding, however, no indications about the presumed superiority of one intervention over the others will be provided to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - Robotic therapy (Experimental): Group A will undergo rehabilitative treatment using Gloreha Sinfonia hand robot, administered by a physical therapist experienced in robotic rehabilitation. The treatment will involve a set of progressively challenging exercises over the course of five weeks (3 sessions per week, each lasting 1 hour). The delivery of the treatment will be conducted in a face-to-face mode.
  Interventions: Device: Robotic therapy (Gloreha Sinfonia system)
- Group B - Occupational Therapy (Experimental): Group B will attend small group occupational therapy treatment (occupational therapist/patient ratio: 1:4). Subjects will attend a rehabilitative intervention lasting a total of 5 weeks, with three sessions per week, each lasting one hour, for a total of 15 hours of treatment.
  Interventions: Other: Occupational therapy
- Group C - Control Group (Active Comparator): Group C (control group) will receive advice from an experienced physiotherapist for a personalized exercise program to be independently carried out at their own residence. The program will focus on the upper limb and will be based on the assessment conducted at baseline.
  Interventions: Behavioral: Control

INTERVENTIONS:
Device: Robotic therapy (Gloreha Sinfonia system) — Group A will receive rehabilitative treatment using the Gloreha Sinfonia system . The treatment regimen spans five weeks and encompasses a progressive series of exercises. Gloreha features an adaptable mechanical design developed for hand rehabilitation. Its activities involve grasping and releasing, facilitated through a lightweight and flexible orthosis. The device, comprising a robotic glove and mechanical arm, enables both finger mobility and upper limb support, facilitating semi-autonomous execution of motor tasks. Gloreha's versatility allows for exercises involving the entire upper limb, including motor-cognitive "serious games" utilizing virtual reality and interaction with real objects. Real-time feedback enhances patient self-assessment. Moreover, the robot incorporates an automated component interfacing with flexion sensors, gauging the patient's autonomous engagement in Occupational Therapy tasks and serious games.
  Arms: Group A - Robotic therapy
Other: Occupational therapy — Occupational Therapy is also recommended in Stroke Rehabilitation Clinical Guidelines. However, its implementation in rehabilitation services in Italy is still limited, presumably due to regulatory factors. For stroke patients, the goal of occupational therapy is to enhance the ability to perform activities of daily living, often focusing on the use of the hand and upper limb in purposeful tasks. Strategies employed by occupational therapists include assessment, treatment, compensation strategies, assistive technologies, and environmental adaptations.
  Occupational therapy appears to enhance performance in activities of daily living and reduce the likelihood of impairment in these abilities, although the evidence is of low quality. There is also limited and moderately quality evidence in the area of occupational therapy for addressing depressive and anxiety symptoms in hospital-based rehabilitation for physical disabilities.
  Arms: Group B - Occupational Therapy
Behavioral: Control — Participants will be provided guidance by a skilled physiotherapist to follow a customized exercise regimen independently within the comfort of their homes. This program will specifically target the upper limb and will be tailored according to the evaluation performed at the initial assessment.
  Arms: Group C - Control Group

SUMMARY:
The functional recovery of the upper limb represents a critical element in post-stroke rehabilitation; hemiplegic/hemiparetic patients who achieve optimal recovery are a minority, and incomplete recovery has relevant consequences both on functioning and on quality of life of those who survive a stroke. The project aims to assess the effects on the functional recovery, with manual dexterity as the primary outcome, of a treatment protocol using an innovative tool (Gloreha Sinfonia) that enables assisted execution of three-dimensional tasks combined with Serious Games for cognitive stimulation, targeting the functional recovery of the upper limb in patients with stroke outcomes at least 6 months after the acute event (chronic phase). Patients with residual dysfunction of the upper limb, at least 6 months after the stroke, will be randomly assigned to the Robotic Rehabilitation group (ROBOT), the Occupational Therapy group (OT), focused on the use of the upper limb in functional tasks (task-oriented training), or the control group (CT - prescription of a home exercise program). Patients in the ROBOT and OT groups will undergo a total treatment period of 5 weeks, with 3 sessions per week lasting 1 hour, for a total of 15 sessions/hours of treatment. Patients assigned to the CT group will undergo an initial functional assessment required for defining the exercise program. All patients will be evaluated at baseline (T0), at a 5-week interval (T1), and 6 months after the end of treatment (T2). Outcome indicators include measures of manual dexterity/upper limb performance, anxiety/depression, cognitive abilities, and patient-perceived outcomes. The analysis of Surface Plasmon Resonance imaging (SPRi) of serum exosome content, detected at T0, T1, and T2, will be correlated with variations in functional measures to verify the hypothesis that induction of neuroplasticity underlies any observed changes. Short- and medium-term effects on functional, psychological outcomes, as well as indicators of neuroinflammation and neural regeneration from serum analysis using innovative SPRi, will be compared among the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. First ischemic or hemorrhagic stroke occurring at least 6 months prior.
2. Persistent motor deficit in the affected upper limb (Motricity Index between 18 and 77).
3. Willingness to participate in the study, with the provision of informed consent.

Exclusion Criteria:

1. Severe spastic hypertonia at the wrist and fingers (Modified Ashworth Scale equal to or greater than 3).
2. Orthopedic, rheumatological, and/or peripheral nervous system disorders affecting the paretic upper limb.
3. Neurodegenerative and neuromuscular disorders.
4. Acute pathologies affecting other body systems.
5. Severe cognitive, language, and behavioral disorders that significantly limit understanding and participation in the planned activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Manual dexterity | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Nine Hole Peg Test (Johansson et al., 2019) - MCID=32s (Sivan et al., 2011); MDC =32,8 sec; Percentage Change=54% (Chen et al., 2009)

SECONDARY OUTCOMES:
Upper limb motor skills | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Wolf Motor Function Test (Wolf et al., 2001) - Minimal Clinically Important Difference (MCID) for Functional Ability: 1.0 points (paretic dominant limb), 1.2 points (paretic non-dominant limb), 17% change (paretic dominant limb), 20% change (paretic non-dominant limb); MCID for Time: -19 seconds, 16% change (paretic dominant limb) (Lang et al., 2008); Minimal Detectable Change (MDC) for timed items: 0.7 seconds; MDC for Functional Ability Scale: 0.1 points (Fritz et al., 2009).
Manual dexterity and activities of daily living abilities | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  ABILHAND questionnaire (Ekstrand et al., 2014) - Minimal Clinically Important Difference (MCID) ranges from 0.26 to 0.35 logits (Wang, 2011).
Anxiety and depression | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Hospital Anxiety and Depression Scale (HADS) (Snaith, 2003) - Minimal Clinically Important Difference (MCID) for Anxiety = 1.96, MCID for Depression = 1.55 (in the context of Cardiovascular Diseases) (Lemay et al., 2018).
Cognitive functioning screening | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Montreal Cognitive Assessment (MOCA) (Shi et al., 2018) - Minimal Detectable Change (MDC) = 3.94 (90% CI), 4.21 (95% CI) - values for the elderly population and geriatric care (Feeney et al., 2016).
Neglect | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Hearts Test (Mancuso et al., 2016)
Health status and quality of life | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Short Form 12 (SF-12) (Gandek et al., 1998) - Minimal Clinically Important Difference (MCID) = 1.8-3.0 units (Fu et al., 2021).
Shoulder/elbow/hand pain | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Numeric Rating Scale (NRS) (Ferreira-Valente et al., 2011) ranging from 0 (no pain) to 10 (worst possible pain)
Participation | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Frenchay Activity Index (FAI) (Antonucci et al., 2022)
Perceived change | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  Seven-level Likert scale (much worse, worse, somewhat worse, about the same, somewhat improved, improved, much improved) (Likert, 1932)
Treatment satisfaction | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  NRS 0-10 (Van Berckel et al., 2016)
Neuroplasticity | At the baseline (beginning of the treatment - T0), at the end of the treatment (T1), and three months after the conclusion of the treatment (T2).
  correlation between outcome measures and variations in surface markers of extracellular vesicles (EVs) as a complex biomarker of neuroplasticity, vascular regeneration, and inflammatory response, assessed through Surface Plasmon Resonance imaging (SPRi)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Cecchi, MD, Principal Investigator — University of Florence; Chiara Castagnoli, PT, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonucci L, Barbato C, Pellicciari L, Paperini A, Hochleitner I, Castagnoli C, Verdesca S, Lucidi G, Marignani S, Pancani S, Basagni B, Macchi C, Cecchi F. Italian translation and cross-cultural validation of an assessment tool for participation in stroke survivors: the Frenchay Activities Index. Neurol Sci. 2022 Jul;43(7):4297-4306. doi: 10.1007/s10072-022-05949-5. Epub 2022 Feb 18. PMID 35179673
- [Background] Aprile I, Germanotta M, Cruciani A, Loreti S, Pecchioli C, Cecchi F, Montesano A, Galeri S, Diverio M, Falsini C, Speranza G, Langone E, Papadopoulou D, Padua L, Carrozza MC; FDG Robotic Rehabilitation Group. Upper Limb Robotic Rehabilitation After Stroke: A Multicenter, Randomized Clinical Trial. J Neurol Phys Ther. 2020 Jan;44(1):3-14. doi: 10.1097/NPT.0000000000000295. PMID 31834217
- [Background] Bennett DA, Krishnamurthi RV, Barker-Collo S, Forouzanfar MH, Naghavi M, Connor M, Lawes CM, Moran AE, Anderson LM, Roth GA, Mensah GA, Ezzati M, Murray CJ, Feigin VL; Global Burden of Diseases, Injuries, and Risk Factors 2010 Study Stroke Expert Group. The global burden of ischemic stroke: findings of the GBD 2010 study. Glob Heart. 2014 Mar;9(1):107-12. doi: 10.1016/j.gheart.2014.01.001. PMID 25432120
- [Background] Bertani R, Melegari C, De Cola MC, Bramanti A, Bramanti P, Calabro RS. Effects of robot-assisted upper limb rehabilitation in stroke patients: a systematic review with meta-analysis. Neurol Sci. 2017 Sep;38(9):1561-1569. doi: 10.1007/s10072-017-2995-5. Epub 2017 May 24. PMID 28540536
- [Background] Cecchi F, Cassio A, Lavezzi S, Scarponi F, Gatta G, Montis A, Bernucci C, Franceschini M, Bargellesi S, Paolucci S, Taricco M. Redefining a minimal assessment protocol for stroke rehabilitation: the new "Protocollo di Minima per l'ICtus" (PMIC2020). Eur J Phys Rehabil Med. 2021 Oct;57(5):669-676. doi: 10.23736/S1973-9087.21.06638-7. Epub 2021 May 27. PMID 34042407
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Background] Chien WT, Chong YY, Tse MK, Chien CW, Cheng HY. Robot-assisted therapy for upper-limb rehabilitation in subacute stroke patients: A systematic review and meta-analysis. Brain Behav. 2020 Aug;10(8):e01742. doi: 10.1002/brb3.1742. Epub 2020 Jun 26. PMID 32592282
- [Background] Cooke SF, Bliss TV. Plasticity in the human central nervous system. Brain. 2006 Jul;129(Pt 7):1659-73. doi: 10.1093/brain/awl082. Epub 2006 May 3. PMID 16672292
- [Background] Crema A, Bassolino M, Guanziroli E, Colombo M, Blanke O, Serino A, Micera S, Molteni F. Neuromuscular electrical stimulation restores upper limb sensory-motor functions and body representations in chronic stroke survivors. Med. 2022 Jan 14;3(1):58-74.e10. doi: 10.1016/j.medj.2021.12.001. Epub 2022 Jan 7. PMID 35590144
- [Background] Dimyan MA, Cohen LG. Neuroplasticity in the context of motor rehabilitation after stroke. Nat Rev Neurol. 2011 Feb;7(2):76-85. doi: 10.1038/nrneurol.2010.200. Epub 2011 Jan 18. PMID 21243015
- [Background] Ekstrand E, Lindgren I, Lexell J, Brogardh C. Test-retest reliability of the ABILHAND questionnaire in persons with chronic stroke. PM R. 2014 Apr;6(4):324-31. doi: 10.1016/j.pmrj.2013.09.015. Epub 2013 Oct 7. PMID 24113290
- [Background] Feeney J, Savva GM, O'Regan C, King-Kallimanis B, Cronin H, Kenny RA. Measurement Error, Reliability, and Minimum Detectable Change in the Mini-Mental State Examination, Montreal Cognitive Assessment, and Color Trails Test among Community Living Middle-Aged and Older Adults. J Alzheimers Dis. 2016 May 31;53(3):1107-14. doi: 10.3233/JAD-160248. PMID 27258421
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Fritz SL, Blanton S, Uswatte G, Taub E, Wolf SL. Minimal detectable change scores for the Wolf Motor Function Test. Neurorehabil Neural Repair. 2009 Sep;23(7):662-7. doi: 10.1177/1545968309335975. Epub 2009 Jun 4. PMID 19498013
- [Background] Fu V, Weatherall M, McNaughton H. Estimating the minimal clinically important difference for the Physical Component Summary of the Short Form 36 for patients with stroke. J Int Med Res. 2021 Dec;49(12):3000605211067902. doi: 10.1177/03000605211067902. PMID 34939887
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186
- [Background] Gualerzi A, Picciolini S, Roda F, Bedoni M. Extracellular Vesicles in Regeneration and Rehabilitation Recovery after Stroke. Biology (Basel). 2021 Aug 30;10(9):843. doi: 10.3390/biology10090843. PMID 34571720
- [Background] Israely S, Leisman G, Carmeli E. Improvement in arm and hand function after a stroke with task-oriented training. BMJ Case Rep. 2017 Mar 17;2017:bcr2017219250. doi: 10.1136/bcr-2017-219250. PMID 28314812
- [Background] Iwamoto Y, Imura T, Suzukawa T, Fukuyama H, Ishii T, Taki S, Imada N, Shibukawa M, Inagawa T, Araki H, Araki O. Combination of Exoskeletal Upper Limb Robot and Occupational Therapy Improve Activities of Daily Living Function in Acute Stroke Patients. J Stroke Cerebrovasc Dis. 2019 Jul;28(7):2018-2025. doi: 10.1016/j.jstrokecerebrovasdis.2019.03.006. Epub 2019 Apr 30. PMID 31047819
- [Background] Johansson GM, Hager CK. A modified standardized nine hole peg test for valid and reliable kinematic assessment of dexterity post-stroke. J Neuroeng Rehabil. 2019 Jan 14;16(1):8. doi: 10.1186/s12984-019-0479-y. PMID 30642350
- [Background] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Background] Lang CE, Edwards DF, Birkenmeier RL, Dromerick AW. Estimating minimal clinically important differences of upper-extremity measures early after stroke. Arch Phys Med Rehabil. 2008 Sep;89(9):1693-700. doi: 10.1016/j.apmr.2008.02.022. PMID 18760153
- [Background] Lang CE, Wagner JM, Edwards DF, Sahrmann SA, Dromerick AW. Recovery of grasp versus reach in people with hemiparesis poststroke. Neurorehabil Neural Repair. 2006 Dec;20(4):444-54. doi: 10.1177/1545968306289299. PMID 17082499
- [Background] Lee HC, Kuo FL, Lin YN, Liou TH, Lin JC, Huang SW. Effects of Robot-Assisted Rehabilitation on Hand Function of People With Stroke: A Randomized, Crossover-Controlled, Assessor-Blinded Study. Am J Occup Ther. 2021 Jan-Feb;75(1):7501205020p1-7501205020p11. doi: 10.5014/ajot.2021.038232. PMID 33399050
- [Background] Legg LA, Lewis SR, Schofield-Robinson OJ, Drummond A, Langhorne P. Occupational therapy for adults with problems in activities of daily living after stroke. Cochrane Database Syst Rev. 2017 Jul 19;7(7):CD003585. doi: 10.1002/14651858.CD003585.pub3. PMID 28721691
- [Background] Lemay KR, Tulloch HE, Pipe AL, Reed JL. Establishing the Minimal Clinically Important Difference for the Hospital Anxiety and Depression Scale in Patients With Cardiovascular Disease. J Cardiopulm Rehabil Prev. 2019 Nov;39(6):E6-E11. doi: 10.1097/HCR.0000000000000379. PMID 30489438
- [Background] Likert R. (1932) Technique for the measure of attitudes Arch. Psycho., Vol. 22 N. 140
- [Background] Mancuso M, Varalta V, Sardella L, Capitani D, Zoccolotti P, Antonucci G; Italian OCS Group. Italian normative data for a stroke specific cognitive screening tool: the Oxford Cognitive Screen (OCS). Neurol Sci. 2016 Oct;37(10):1713-21. doi: 10.1007/s10072-016-2650-6. Epub 2016 Jul 9. PMID 27395388
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2015 Nov 7;2015(11):CD006876. doi: 10.1002/14651858.CD006876.pub4. PMID 26559225
- [Background] Mehrholz J, Pollock A, Pohl M, Kugler J, Elsner B. Systematic review with network meta-analysis of randomized controlled trials of robotic-assisted arm training for improving activities of daily living and upper limb function after stroke. J Neuroeng Rehabil. 2020 Jun 30;17(1):83. doi: 10.1186/s12984-020-00715-0. PMID 32605587
- [Background] Meyer S, Karttunen AH, Thijs V, Feys H, Verheyden G. How do somatosensory deficits in the arm and hand relate to upper limb impairment, activity, and participation problems after stroke? A systematic review. Phys Ther. 2014 Sep;94(9):1220-31. doi: 10.2522/ptj.20130271. Epub 2014 Apr 24. PMID 24764072
- [Background] Pisegna J, Anderson S, Krok-Schoen JL. Occupational Therapy Interventions to Address Depressive and Anxiety Symptoms in the Physical Disability Inpatient Rehabilitation Setting: A Systematic Review. Am J Occup Ther. 2022 Jan 1;76(1):7601180110. doi: 10.5014/ajot.2022.049068. PMID 35037944
- [Background] Ramos-Murguialday A, Schurholz M, Caggiano V, Wildgruber M, Caria A, Hammer EM, Halder S, Birbaumer N. Proprioceptive feedback and brain computer interface (BCI) based neuroprostheses. PLoS One. 2012;7(10):e47048. doi: 10.1371/journal.pone.0047048. Epub 2012 Oct 5. PMID 23071707
- [Background] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Background] Shi D, Chen X, Li Z. Diagnostic test accuracy of the Montreal Cognitive Assessment in the detection of post-stroke cognitive impairment under different stages and cutoffs: a systematic review and meta-analysis. Neurol Sci. 2018 Apr;39(4):705-716. doi: 10.1007/s10072-018-3254-0. Epub 2018 Feb 9. PMID 29427168
- [Background] Sivan M, O'Connor RJ, Makower S, Levesley M, Bhakta B. Systematic review of outcome measures used in the evaluation of robot-assisted upper limb exercise in stroke. J Rehabil Med. 2011 Feb;43(3):181-9. doi: 10.2340/16501977-0674. PMID 21305232
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Sommerfeld DK, von Arbin MH. The impact of somatosensory function on activity performance and length of hospital stay in geriatric patients with stroke. Clin Rehabil. 2004 Mar;18(2):149-55. doi: 10.1191/0269215504cr710oa. PMID 15053123
- [Background] Stinear CM, Lang CE, Zeiler S, Byblow WD. Advances and challenges in stroke rehabilitation. Lancet Neurol. 2020 Apr;19(4):348-360. doi: 10.1016/S1474-4422(19)30415-6. Epub 2020 Jan 28. PMID 32004440
- [Background] Turner DL, Ramos-Murguialday A, Birbaumer N, Hoffmann U, Luft A. Neurophysiology of robot-mediated training and therapy: a perspective for future use in clinical populations. Front Neurol. 2013 Nov 13;4:184. doi: 10.3389/fneur.2013.00184. PMID 24312073
- [Background] Tyson SF, Hanley M, Chillala J, Selley AB, Tallis RC. Sensory loss in hospital-admitted people with stroke: characteristics, associated factors, and relationship with function. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):166-72. doi: 10.1177/1545968307305523. Epub 2007 Aug 8. PMID 17687023
- [Background] van Berckel MM, Bosma NH, Hageman MG, Ring D, Vranceanu AM. The Correlation Between a Numerical Rating Scale of Patient Satisfaction With Current Management of an Upper Extremity Disorder and a General Measure of Satisfaction With the Medical Visit. Hand (N Y). 2017 Mar;12(2):202-206. doi: 10.1177/1558944716662019. Epub 2016 Aug 19. PMID 28344535
- [Background] Vanoglio F, Bernocchi P, Mule C, Garofali F, Mora C, Taveggia G, Scalvini S, Luisa A. Feasibility and efficacy of a robotic device for hand rehabilitation in hemiplegic stroke patients: a randomized pilot controlled study. Clin Rehabil. 2017 Mar;31(3):351-360. doi: 10.1177/0269215516642606. Epub 2016 Jul 10. PMID 27056250
- [Background] Villafane JH, Taveggia G, Galeri S, Bissolotti L, Mulle C, Imperio G, Valdes K, Borboni A, Negrini S. Efficacy of Short-Term Robot-Assisted Rehabilitation in Patients With Hand Paralysis After Stroke: A Randomized Clinical Trial. Hand (N Y). 2018 Jan;13(1):95-102. doi: 10.1177/1558944717692096. Epub 2017 Feb 16. PMID 28719996
- [Background] Wang TN, Lin KC, Wu CY, Chung CY, Pei YC, Teng YK. Validity, responsiveness, and clinically important difference of the ABILHAND questionnaire in patients with stroke. Arch Phys Med Rehabil. 2011 Jul;92(7):1086-91. doi: 10.1016/j.apmr.2011.01.020. PMID 21704789
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Wolf SL, Catlin PA, Ellis M, Archer AL, Morgan B, Piacentino A. Assessing Wolf motor function test as outcome measure for research in patients after stroke. Stroke. 2001 Jul;32(7):1635-9. doi: 10.1161/01.str.32.7.1635. PMID 11441212